CLINICAL TRIAL: NCT02289560
Title: A Continued Access Study to Evaluate the Effectiveness and Safety of ExAblate Transcranial MRgFUS Thalamotomy Treatment of Medication Refractory Essential Tremor Subjects
Brief Title: Continued Access Protocol: ExAblate Transcranial MR Guided Focused Ultrasound for the Treatment of Essential Tremors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET002CA
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcranial ExAblate (Experimental): Transcranial ExAblate
  Interventions: Device: Transcranial ExAblate

INTERVENTIONS:
Device: Transcranial ExAblate — Transcranial ExAblate
  Other Names: ExAblate; TcMRgFUS; Thalamotomy

SUMMARY:
The objective of this prospective, multi site, single-arm study is to capture the efficacy of treatment using the ExAblate Transcranial System and to further demonstrate safety in medication-refractory tremor in patients with essential tremor (ET).

DETAILED DESCRIPTION:
This study is evaluating a new technique for performing Thalamotomy for tremor control. While current techniques have possible invasive or radiation effects, the use of ExAblate if totally non-invasive and without any radiation. After informed consent and screening, eligible subjects will be undergo an ExAblate treatment. All subjects will be followed at 1 day, 1 week, 1, 3, 6 and 12 months and for up to 5 years as directed by their doctor.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 22 years and older
* Subjects who are able and willing to give informed consent and able to attend all study visits
* Subjects with a diagnosis of Essential Tremor as confirmed from clinical history and examination by a neurologist or neurosurgeon specialized in movement disorder
* Subject exhibits a significant disability from their ET despite medical treatment
* Subjects should be on a stable dose of all ET medications for 30 days prior to study entry
* Subject is able to communicate sensations during the ExAblate Transcranial procedure

Exclusion Criteria:

* Subjects with unstable cardiac status
* Severe hypertension
* Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Known intolerance or allergies to the MRI contrast agent including advanced kidney disease or severely impaired renal function
* Significant claustrophobia that cannot be managed with mild medication
* Current medical condition resulting in abnormal bleeding and/or coagulopathy
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage
* History of intracranial hemorrhage
* History of multiple strokes, or a stroke within past 6 months
* Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment
* Are participating or have participated in another clinical trial in the last 30 days
* Subjects unable to communicate with the investigator and staff
* Subjects with a history of seizures within the past year
* Subjects with brain tumors

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Stanford University Medical Center, Stanford, California
  - University of Maryland Medical System, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - The Ohio State Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- Available data/document: Clinical Study Report — https://www.accessdata.fda.gov/cdrh_docs/pdf15/p150038c.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Exablate: Transcranial Exablate: This was a single-arm study with no proposed hypothesis. All subjects were treated with unilateral transcranial Exablate for essential tremor.
Period: Overall Study
Arm/Group | Transcranial Exablate
Started | 61
Completed | 26
Not Completed | 35
Not completed — Lost to Follow-up | 6
Not completed — Alternative Treatment | 4
Not completed — Inadequate Treatment | 2
Not completed — Withdrawal by Subject | 23

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial ExAblate
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Birth date was not reported for three subjects
  years
    number analyzed (Participants) | 58
    (all) | 69.5 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57
  Hispanic | 0
  Black | 0
  Asian | 3
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 61
Family History of Essential Tremor [Count of Participants; unit: Participants]
  Yes | 45
  No | 15
  Unknown | 1
Years of Essential Tremor History [Mean (Standard Deviation); unit: years] — Population: Family history of essential tremor was not reported for one subject out of 61. Thus, n=60 subjects were available for summary statistical analysis.
  years
    number analyzed (Participants) | 60
    (all) | 19.5 (14.2)
Skull Density Ratio [Mean (Standard Deviation); unit: Ratio] — Population: SDR was not reported for four subjects
  Ratio
    number analyzed (Participants) | 57
    (all) | 0.54 (0.10)
Clinical Rating Scale for Tremor - Tremor Motor Score [Mean (Standard Deviation); unit: Score on a Scale] — Baseline sum of upper extremity Tremor-Motor scores for the treated side from the Clinical Rating Scale for Tremor (CRST) Part A and Part B averaged across subjects. This measure of upper extremity tremor ranges from 0-32 with high scores being worse. Lower scores are better than higher scores.
  Score on a Scale | 19.0 (4.9)
Quality of Life for Essential Tremor (QUEST) Summary of Dimensions TOTAL Score [Mean (Standard Deviation); unit: Score on a scale] — Measure Description: Baseline Quality of Life for Essential Tremor (QUEST) TOTAL is the mean of five QUEST dimensions each as a percent of the total possible. The QUEST is a 30-item assessment with each item scored 0-4 (total min - max is 0 - 120). For each subject, each of the 5 QUEST dimension scores is a percentage (100%-0%) of total possible for each dimension. The QUEST summary of dimensions total is a mean of the five dimension scores. Lower QUEST scores are better than higher scores.
  Score on a scale | 42.9 (17.4)
CRST Part C Functional Disabilities Score [Mean (Standard Deviation); unit: Score on a Scale] — Baseline Clinical Rating Scale for Tremor (CRST) Part C is a measure of functional disability due to tremor. The Clinical Rating Scale for Tremor Part C consists of 8 items each scored from 0 to 4. Thus, the total score summed ranges from 0 to 32 (average, 0-4) and provides an overall assessment of activities of daily living. Low scores on the Clinical Rating Scale for Tremor (CRST) Part C are better. Low scores show improvement in functional disabilities compared to higher scores.
  Score on a Scale | 16.7 (4.87)

OUTCOME MEASURES:

1. Primary Outcome: Number of Device and Procedure Related Adverse Events.
Description: The cumulative sum of adverse events was followed through Year 5 of the study.
Time Frame: 5 Years post treatment
Population: Adverse Events and Serious Adverse Events are Presented in Adverse Events Section
Measure: Number; unit: Number of adverse events
Arm/Group | Transcranial ExAblate
Number analyzed (Participants) | 61
Number of adverse events | 121

2. Secondary Outcome: Tremor Motor Score - Clinical Rating Scale for Tremor (CRST) Part A (Upper Extremity) + Part B Scores Summed
Description: Sum of baseline and follow-up in upper extremity Tremor-Motor scores for the treated side is a sub-scale of Clinical Rating Scale for Tremor (CRST) Part A and Part B sum that was used to measure treated-side upper extremity tremor changes over time. Tremor-motor scores range from 0-32 points. Individual subject's scores at Baseline and Follow Up were calculated at baseline and follow-up visits averaged across subjects. Low scores are better (show improvement).
Time Frame: Baseline, 3 Months, 6 Months, 12 Months, 2, 3, 4, 5 Years post treatment
Population: Sixty-one subjects were treated. Follow-up measures included all subjects completing the assessments. Subjects withdrawn from the study, missed visits, or missed assessments were not imputed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Transcranial Exablate
Number analyzed (Participants) | 61
score on a scale
  Baseline | 19.0 [17.80 to 20.26]
  Month 3 Follow Up: number analyzed (Participants) | 55
  Month 3 Follow Up | 6.3 [4.88 to 7.70]
  Month 6 Follow Up: number analyzed (Participants) | 55
  Month 6 Follow Up | 7.0 [5.43 to 8.57]
  Month 12 Follow Up: number analyzed (Participants) | 53
  Month 12 Follow Up | 7.4 [5.81 to 8.90]
  2 Year Follow Up: number analyzed (Participants) | 45
  2 Year Follow Up | 7.3 [5.80 to 8.78]
  3 Year Follow Up: number analyzed (Participants) | 35
  3 Year Follow Up | 7.3 [5.66 to 8.91]
  4 Year Follow Up: number analyzed (Participants) | 31
  4 Year Follow Up | 7.9 [5.92 to 9.95]
  5 Year Follow Up: number analyzed (Participants) | 23
  5 Year Follow Up | 9.2 [6.70 to 11.73]

3. Secondary Outcome: Clinical Rating Scale for Tremor (CRST Part A) Posture Score Change From Baseline
Description: The Posture Score is a sub-Score of the Clinical Rating Scale for Tremor CRST Part A - Posture (Treated Side Upper Extremity Posture Score). The minimum-maximum average score range is 0-4 and higher scores indicate worse outcomes.
Time Frame: Baseline, 3 Months, 6 Months, 12 Months, 2, 3, 4, 5 Years post treatment
Population: Sixty-one subjects were treated. Follow-up measures included all subjects completing the assessments. Subjects withdrawn from the study, missed visits, or missed assessments were included. Missing scores were not imputed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Transcranial Exablate
Number analyzed (Participants) | 61
score on a scale
  Baseline | 2.8 [2.54 to 3.01]
  Month 3 Follow Up: number analyzed (Participants) | 56
  Month 3 Follow Up | 0.7 [0.44 to 0.88]
  Month 6 Follow Up: number analyzed (Participants) | 56
  Month 6 Follow Up | 0.8 [0.55 to 1.06]
  Month 12 Follow Up: number analyzed (Participants) | 53
  Month 12 Follow Up | 0.7 [0.46 to 0.90]
  Year 2 Follow Up: number analyzed (Participants) | 45
  Year 2 Follow Up | 0.5 [0.29 to 0.69]
  Year 3 Follow Up: number analyzed (Participants) | 36
  Year 3 Follow Up | 0.6 [0.39 to 0.78]
  Year 4 Follow Up: number analyzed (Participants) | 32
  Year 4 Follow Up | 0.7 [0.38 to 0.93]
  Year 5 Follow Up: number analyzed (Participants) | 23
  Year 5 Follow Up | 0.9 [0.51 to 1.32]

4. Secondary Outcome: Clinical Rating Scale for Tremor Part C - Activities of Daily Living.
Description: Subject daily functionalities as measured by Clinical Rating Scale for Tremor Part C, CRST Part-C (subscales). CRST Part-C is an 8-item score with a minimum-maximum range of 0-32. Higher scores mean worse outcomes.
Time Frame: Baseline, 3 Months, 6 Months, 12 Months, 2, 3, 4, 5 Years post treatment
Population: The population includes all Exablate-treated subjects. Sample size at each visit includes all subjects excluding those that withdrew consent or missed the visit assessment. Missing scores were not imputed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Transcranial Exablate
Number analyzed (Participants) | 61
score on a scale
  Baseline | 16.7 [15.47 to 17.91]
  Month 3: number analyzed (Participants) | 56
  Month 3 | 3.5 [2.47 to 4.46]
  Month 6: number analyzed (Participants) | 56
  Month 6 | 3.8 [2.41 to 5.09]
  Month 12: number analyzed (Participants) | 53
  Month 12 | 5.8 [4.20 to 7.46]
  2 Year Follow Up: number analyzed (Participants) | 45
  2 Year Follow Up | 6.1 [4.39 to 7.74]
  3 Year Follow Up: number analyzed (Participants) | 35
  3 Year Follow Up | 8.3 [5.95 to 10.62]
  4 Year Follow Up: number analyzed (Participants) | 32
  4 Year Follow Up | 8.4 [6.12 to 10.70]
  5 Year Follow Up: number analyzed (Participants) | 23
  5 Year Follow Up | 10.4 [7.26 to 13.52]

5. Secondary Outcome: Quality of Life in Essential Tremor Total (QUEST)
Description: The QUEST Summary Total was used to assess quality of life changes over time in tremor patients. The QUEST consists of five dimensions for each subject converted to a percent of the total (0-100%). The summary total is the average of the five dimensions. Low Total scores are better.
Time Frame: Baseline, 3 Months, 6 Months, 12 Months, 2, 3, 4, 5 Years post treatment
Population: The population includes all Exablate treated subjects except for those withdrawing consent or missing the assessment. Missing scores were not imputed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Transcranial Exablate
Number analyzed (Participants) | 61
score on a scale
  Baseline | 42.9 [38.51 to 47.25]
  Month 3: number analyzed (Participants) | 56
  Month 3 | 17.8 [12.81 to 22.71]
  Month 6: number analyzed (Participants) | 57
  Month 6 | 18.6 [13.64 to 23.52]
  Month 12: number analyzed (Participants) | 53
  Month 12 | 19.60 [14.22 to 24.88]
  Year 2 Follow Up: number analyzed (Participants) | 45
  Year 2 Follow Up | 21.0 [15.24 to 26.84]
  Year 3 Follow Up: number analyzed (Participants) | 35
  Year 3 Follow Up | 24.0 [17.75 to 30.17]
  Year 4 Follow Up: number analyzed (Participants) | 31
  Year 4 Follow Up | 22.5 [15.59 to 29.44]
  Year 5 Follow Up: number analyzed (Participants) | 22
  Year 5 Follow Up | 25.1 [15.98 to 34.30]

ADVERSE EVENTS:
Time Frame: Intraprocedural cumulative through 5 Years
Description: Intraprocedural, at ea. follow-up visit (1 Month, 3 Month, 6 Month, 12 Month and annually through Year 5
Arm/Group | Transcranial Exablate
All-Cause Mortality (participants affected / at risk) | 3/61
Serious Adverse Events (participants affected / at risk) | 2/61
Other Adverse Events (participants affected / at risk) | 52/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Exablate (N=61)
Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) (Nervous system disorders) | 1 (1) — Developed gait imbalance and dysmetria of the upper extremities and right lower extremity which worsened over time and was determined to be related to the thalamotomy procedure.
Myocardial Infarction. (Cardiac disorders) | 1 (1) — The subject was treated for procedure-related myocardial infarction and subsequently did well with tremor relief and no further cardiac issues.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Exablate (N=61)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Lethargy (General disorders) | 1 (1)
IV site infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Imbalance (Nervous system disorders) | 1 (1)
Numbness/Tingling (Surgical and medical procedures) | 1 (1)
Headache (Surgical and medical procedures) | 5 (5)
Jaw pain (Surgical and medical procedures) | 1 (1)
Edema (Surgical and medical procedures) | 1 (1)
Imabalance (Ear and labyrinth disorders) | 9 (9)
Dysgnathia (Surgical and medical procedures) | 2 (2)
Vision problem (Eye disorders) | 2 (2)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemi-body muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Imbalance (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myoclonus (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 10 (10)
Dysarthria (Nervous system disorders) | 7 (7)
Dysgeusia (Nervous system disorders) | 6 (6)
Dysmetria (Nervous system disorders) | 7 (9)
Gait disturbance (Nervous system disorders) | 9 (9)
Imbalance (Nervous system disorders) | 11 (11)
Numbness/Tingling (Nervous system disorders) | 20 (29)
Slurred speech (Nervous system disorders) | 1 (1)
Unclear thinking (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT02289560/Prot_SAP_000.pdf